CLINICAL TRIAL: NCT06767254
Title: A Machine Learning Approach to Connect Multiple Myeloma Complexity to Early Disease Recurrence
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: AIMMer; PNRR-TR1-2023-12378246 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-01-02; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, national, multicenter prospective non-profit observational study aiming at improving the accuracy of risk prediction in multiple myeloma (MM) by applying machine-learning tools for data processing to develop model(s) predicting response to therapy and the probability of early relapse for MM patients.

DETAILED DESCRIPTION:
Improvements in the therapy of MM have prompted the achievement of very deep clinical responses, with significantly improved outcomes and survival [2]. However, despite significant therapeutic progress, MM remains a challenge, due to the composite pathogenesis and intricate networks of different interacting factors. As a result, a relatively high proportion of NDMM patients across the different therapeutic strategies have a higher risk of disease progression and worse outcomes, independently of the anti-MM regimen received. These patients currently represent un unmet clinical need, with consequent challenges in the management of the disease and identify these patients upfront is an important goal in MM.

At present, risk stratification scores rely on a limited set of clinical and biological variables, not always sufficient to identify patients at a high risk of early disease progression or relapse (i.e., within 12 months from start of first-line therapy). Recently, AI tools have been explored to improve the accuracy of risk prediction, showing that high-risk diseases might be upfront recognized, based on tumor and immune biomarkers [3-4].

By applying Machine Learning (ML) tools for data processing, clinical, genomic, and imaging data from MM patients will be integrated and employed in models aimed at improving the accuracy of MM risk prediction. In this way, ML models will aggregate all tumor- and microenvironment-related information obtained by high-throughput technologies and omics approaches to identify and describe clusters of MM patients that best correlate with the achievement of early progression.

Overall, this study will identify new knowledge to support clinical research and decision-making in MM: precise up-front stratification of patients, based on the whole landscape of MM-related features, could improve understanding of MM individual risk. Results from this study will have an impact on the possibility to access personalized treatment, with predictable overall repercussion on the effective management of MM patients and savings for the National Health System.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed Informed Consent form for study participation and personal data processing
* Diagnosis of active multiple myeloma

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be adult patients with newly diagnosed (ND) multiple myeloma.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 12 months after the start of anti-MM therapy
  Overall Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Elena Zamagni, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (4):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST IRCCS, Meldola, Forlì-Cesena
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - ARNAS "G. Brotzu" di Cagliari, Cagliari
  - Azienda Ospedaliera Universitaria Federico II, Napoli

IPD SHARING:
Plan to Share IPD: No